CLINICAL TRIAL: NCT01817829
Title: Oral Paracetamol as Preemptive Analgesia for Labor Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPPALP; Personal (Other: Ain Shams)
Record Dates: First submitted 2013-02-04; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- paracetamol (Active Comparator): paracetamol 2 tablets1000mg PO.
  Interventions: Drug: paracetamol
- placebo (Placebo Comparator): placebo 2 tablets containing Starch PO
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paracetamol — 500 mg oral tablet
  Arms: paracetamol
Drug: placebo
  Arms: placebo

SUMMARY:
It is a double blinded randomized control trial assessing the use of Oral paracetamol in managing the intrapartum pain.

DETAILED DESCRIPTION:
It is a double blinded randomized control trial comparing the use of Oral paracetamol to placebo in managing the intrapartum pain.

ELIGIBILITY:
Inclusion Criteria:

* primigravida
* The gestational age between 37- 42 weeks
* Not seeking analgesia
* Singleton pregnancy
* vertex
* Spontaneous onset of labour
* 1st stage of labour (less than 5 cm)

Exclusion Criteria:

* Extreme of age (below18-above 40)
* Multiparous
* Multiple gestation
* Malpresentation
* Congenital or acquired pelvic abnormalities(eg. Poliomyelitis)
* Any medical disorder with pregnancy
* Induction of labour
* Advanced 1st stage > 5 cm
* Use of any other kind of analgesia before recruitment in the study
* Scared uterus
* Fetal distress

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | intrapartum
  To document the efficacy of oral paracetamol, in pregnant women in labor, as demonstrated by the degree of pain relief and need for additional analgesia during the labor process and the early postpartum period.

SECONDARY OUTCOMES:
Safety | Start of medication till 24 hours postpartum
  To document safety and evaluate adverse events recorded during the study either maternal or fetal.
Duration of labor | Start of medication till delivery of fetus.
  To assess the effect of the duration of labor.